CLINICAL TRIAL: NCT00487370
Title: Extraarticular Gold Implantation for Treatment of Knee Osteoarthritis.
Brief Title: Implantation of Gold Beads to Relieve Discomfort From Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KN1996
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2007-06-18 (Estimated); Status verified 2007-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Acupuncture; Gold implantation; Osteoarthritis; Knee osteoarthritis; Double-blind, randomized controlled trial; Intervention; Family practice
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Implantation of gold beads around a knee through needles
Procedure: Sham implantation: Insertion of needles around a knee

SUMMARY:
The purpose of this study is to determine whether implanting gold beads extraarticularly in five acupuncture-points around a knee improves pain, stiffness and function in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most common diagnoses made in general practice and among the most common causes of disability in older people. Acupuncture is a well-founded supplement or alternative to pharmacological and surgical treatment methods. The improvement is, however, often brief, so to preserve the initial effect the acupuncture has to be repeated at regular intervals.

In veterinarian medicine implantation of gold-beads in acupuncture-points around a joint has been used mostly in dogs for at least 30 years in the treatment of OA. The effect measured on eating pattern, physical activity and signs of pain last for several years. It may be hypothesized that implanting gold in acupuncture points acts as a continuous acupuncture stimulation.

The purpose of this one year randomised, controlled trial of middle-aged and elderly patients is to examine the effect of implanting gold beads extraarticularly in five acupuncture-points around a knee with OA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Clinically diagnosed and radiologically verified knee osteoarthritis (OA)
* Pain and stiffness derived from OA lasting for more than one year

Exclusion Criteria:

* Previous knee trauma (OA following previous meniscectomy is included)
* Other rheumatologic conditions like rheumatoid arthritis or fibromyalgia
* Pronounced hip OA
* Severe somatic or mental illnesses
* Dementia
* Alcohol or drug abuse
* Pregnancy
* Anticoagulant treatment
* Corticosteroid treatment during the last 3 months
* Allergy to chlorhexidine or local anaesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 1997-03; Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Pain from the knee osteoarthritis is evaluated by the patient with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). | 0, 1, 3, 6, 9, and 12 months
Stiffness is evaluated with the WOMAC questionnaire. | 0, 1, 3, 6, 9, and 12 months
Function is evaluated with the WOMAC questionnaire. | 0, 1, 3, 6, 9, and 12 months
The same orthopaedic surgeon assesses the patients knee score using the Knee Society Clinical Rating System. | 0, 6, and 12 months
The same orthopaedic surgeon assesses the patients function score using the Knee Society Clinical Rating System. | 0, 6, and 12 months

SECONDARY OUTCOMES:
The effect of the initial screening by conventional acupuncture - in relation to the five primary outcome measures. | 2 months before randomisation
Side-effects and discomfort from the implantation, primarily whether the implanted gold beads will migrate during the study period. | The entire study period
The time from implantation until the effect possibly sets in. | The entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nejrup, MD, Principal Investigator — General practice, Dronninggårds Alle 2 B, DK-2840 Holte, Denmark
Locations (1):
- General practice, Holte, Denmark